CLINICAL TRIAL: NCT03839589
Title: Adaptation and Implementation of a Mindfulness Intervention Among a Hispanic Immigrant Population in St. Louis
Brief Title: MBSR in a Hispanic Immigrant Population in St. Louis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Diana Parra Perez, Assistant Profesor, Washington University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 212832
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Mindfulness; Emotional Well-being
Keywords: Hispanics; Mindfulness; Emotional well-being

STUDY DESIGN:
Intervention Model Description: We will use a wait-listed design versus a standard parallel group RCT because the wait-listed design allows all participants to (eventually) receive the intervention, and maximizes the overall amount of information obtained. A wait-listed design has been previously used by the primary mentor of this award, Dr. Lenze; successfully increasing recruitment, retention and adherence of the intervention and control groups. This design also allows us to get participant feedback in the whole sample and get preliminary estimates of outcomes, which will be crucial to inform the proposed R01 to be submitted by year 4 of the current award.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to the intervention assignment. Within the resources available to this study, intervention staff will not be engaged in evaluating participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSR-A (Experimental): Intervention Mindfulness Condition: MBSR is a structured intervention delivered through an 8-week course. Mindful breathing, awareness, walking, and attention are core activities taught and practiced during and outside of the course.
  Interventions: Behavioral: Mindfulness Based Stress Reduction Adapated (MBSR-A)
- Wait-listed MBSR-A (Placebo Comparator): The MBSR-A Wait-listed group: This wait-listed group will be followed with the same outcome assessments as the MBSR- A immediate group but will receive no intervention until after outcomes from group 1 are collected at 3 months, when they will also receive the MBSR-A
  Interventions: Behavioral: Mindfulness Based Stress Reduction Adapated (MBSR-A)

INTERVENTIONS:
Behavioral: Mindfulness Based Stress Reduction Adapated (MBSR-A) — Mindfulness-based stress reduction (MBSR) is a group-based intervention developed in 1979 by Dr. Jon Kabat-Zinn to provide mindfulness training in order to decrease stress and improve overall well-being. MBSR has been shown to be effective for a series of patient outcomes including depression, anxiety disorders, sleep disorders, and chronic pain management. MBSR is a structured intervention delivered through an 8-week course of up to 30 participants who meet for 2.5 hours per week.

SUMMARY:
Hispanics are the largest ethnic group in the US as well as the fastest growing. Yet, despite being such a large population group, Hispanics are under-studied and under-represented in most studies of health, psychological well-being, and mind-body interventions. For many Hispanic immigrants, life in the U.S. carries multiple socio-economic stressors, which places them at higher risk for depression and other poor health-related quality of life outcomes. Mindfulness-based stress reduction (MBSR) is a group-based training shown to reduce stress and improve overall well-being. There is a quality gap about adaptation and implementation of MBSR programs in community settings and among Hispanic immigrants. This K23 seeks to adapt and test the implementation of an MBSR intervention among under-resourced Hispanic immigrants in St. Louis guided by methods and frameworks from the field of dissemination and implementation (D&I) science as applied to community settings. Implementation research of mindfulness-based interventions among Hispanic immigrant populations is justifiable under several conditions, including ineffective clinical engagement with this population, risk or resilience factors that are unique to the Hispanic community, and lack of cultural relevance of many evidence-based MBIs.

DETAILED DESCRIPTION:
This career development award will establish Dr. Parra as a clinical translational investigator focused on mind-body interventions for Hispanic immigrant populations. This K23 award will provide her the support needed to develop expertise in 3 areas: (1) Training to conduct well designed randomized clinical trials; (2) Dissemination and Implementation (D&I) science; and (3) Mindfulness research. To achieve these goals, Dr. Parra has assembled an expert multidisciplinary team in clinical research, D&I, and mindfulness. Her primary mentor, Dr. Eric Lenze, has extensive experience in conducting randomized clinical trials and mentoring junior faculty to become independent investigators. Her secondary mentor, Dr. Ross Brownson, is an internationally recognized and leading expert in D&I science. Her scientific collaborators and advisors include Dr. Douglas Ziedonis, a leading expert in mindfulness clinical research and Dr. Tod Braver, a mindfulness research expert. Dr. Parra will also benefit from the expertise of two renowned researchers in D&I science in the areas of intervention adaptation (Dr. Ana Baumann) and measuring implementation and feasibility outcomes (Dr. Rachel Tabak), as well as the experience from a senior MBSR expert (Dr. Jeannie Kloeckner), and an expert on mental health interventions for Hispanic populations (Dr. Patricia Cavazos-Rehg). Hispanics are the largest and fastest-growing ethnic group in the US, currently representing 14 percent of the population. Despite this, Hispanics are seldom represented in research studies and health promoting programs, in part due to a lack of cultural appropriateness by researchers and low levels of trust of the research community by many Hispanics. Using D&I frameworks and methods, Dr. Parra will adapt a Mindfulness Based Stress Reduction intervention (MBSR-A) among under-resourced Hispanic immigrants in St. Louis (Aim 1). Dr. Parra will also conduct a pilot feasibility RCT trial among 60 Hispanic immigrants (Aim 2) to test and measure implementation outcomes including acceptability, appropriateness and feasibility. This research plan leverages existing institutional resources at Washington University in St. Louis (WU), including the Healthy Mind Lab from Dr. Lenze, Dr. Brownson's D&I center, as well as Dr. Lenze's and Dr. Braver's NIH-funded mindfulness research groups. Finally, this training and research will form the basis for an R01 application to further study the adoption, implementation and effectiveness of a Mindfulness intervention in under-resourced Hispanic immigrant populations.

ELIGIBILITY:
Inclusion Criteria:

* Non-institutionalized adult Hispanic men and women attending community centers in St. Louis that serve the immigrant population, under resourced (those earning less than twice the federal poverty line)42, less than five years of having immigrated to the United States, low to normal English literacy, and no history of cognitive or physical disability that would prevent participation. Participants must not be currently involved in any other type of mind-body intervention.

Exclusion Criteria:

* participants with a history of cognitive or physical disability that would prevent participation.
* participants currently involved in any other type of mind-body intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-11-26 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

PRIMARY OUTCOMES:
Emotional well-being | 6 months
  We will use the NIH Toolbox Emotion Battery (NIHTB-EB) for adults. The NIHTB-EB is a computerized assessment of emotions with 17 scales and four theoretically driven subdomains (negative affect, psychological well-being, stress and self-efficacy, and social relationships) with established psychometric properties. The battery takes 20 to 30 minutes to complete, and is self-administered. Each item is assessed on a 5 to 7 point Likert scale (ranging from "not at all" to "very much") and scored using item response theory (IRT) that generates a theta score. Spanish versions of the questionnaire are available and have been tested for psychometric properties in Hispanic populations, showing strong reliability and validity.

SECONDARY OUTCOMES:
Mindfulness | 6 months
  The Mindfulness Attention Awareness Scale (MAAS) will be used to evaluate quality of consciousness and well-being associated with increased self-awareness.61 The 15-item measure uses a 6-point scale to ask participants how often they experience mindful thinking and awareness, with response options ranging from "1-Almost always" to "6-Almost never." An average is taken of the 15 responses for a total possible score range from 1 - 6 with higher scores indicating greater mindful awareness. A translated version of this scale has been previously used in Spanish-speaking community settings and tested for psychometric properties showing high levels of reliability and validity.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Medical information/PHI that is collected for recruitment purposes will be kept on a secured server and/or protected under the 2-key lock concept. Collected information will be de-identified and stored on a secure network drive. The participant will have the right to refuse any study tests. All the tests performed will help us better understand the effect of a mindfulness based stress reduction intervention on emotional well-being and will not invade the privacy of the participants. We do no plan to share the infiormation from the participants with other researchers.